CLINICAL TRIAL: NCT04086615
Title: Trial of Neurostimulation and Blood Flow Restriction for PFPS in Active Duty
Acronym: BFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Blanchfield Army Community Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N19-B01
Record Dates: First submitted 2019-09-03; First posted 2019-09-11 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2021-09

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: 84 (anticipated) participants will be assigned to one of two parallel groups. Sample size was determined using 1) an alpha level of 0.05 and power of 0.80; 2) review of PFPS literature and data from pilot work; and 3) calculation of effect sizes for key variables from previous studies that addressed the Specific Aims.
  For the primary outcome variable of strength, the sample size calculated was 35 subjects per groups (70 total subjects) with an effect size of 0.52. For the outcomes measures of function, mobility and pain, assuming that standard errors will be similar to those observed in our previous work, the sample size of 35 per group is sufficient to detect the expected mean changes. To account for dropouts, the investigators inflated the sample size by 20%, for a total of 42 subjects per group and a total sample size of 84.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- NMES and exercise supplemented with high BFR (Experimental): All participants receive a standard exercise rehabilitation protocol for PFPS to be performed singularly at home/work, synchronously with NMES and concurrently with NMES/BFR in-clinic. The PFPS exercises teach muscle strengthening exercises and self-management strategies to prevent recurrence. Participants will receive a portable battery-operated device, KneeHAB® XP (Bio-Medical Research, Galway, Ireland) with the thigh garment. NMES training will consist of 20-minute stimulation sessions performed concurrently with the exercise program.
  For the BFR training, the automatic Delfi's PTS Personalized Tourniquet System for Blood Flow Restriction (Delfi Medical, Vancouver, BC, Canada) with variable contour nylon cuff (11.5 cm × 86 cm, 2.5 mm thick) will be used. The Delfi PTS system automatically adjusts pressure around the set occlusion pressure. The High BFR group will have the pressure set at 80% of limb occlusion pressure.
  Interventions: Device: NMES and exercise supplemented with high BFR
- NMES and exercise supplemented with low BFR (Sham Comparator): All participants receive a standard exercise rehabilitation protocol for PFPS to be performed singularly at home/work, synchronously with NMES and concurrently with NMES/BFR in-clinic. The PFPS exercises teach muscle strengthening exercises and self-management strategies to prevent recurrence. Participants will receive a portable battery-operated device, KneeHAB® XP (Bio-Medical Research, Galway, Ireland) with the thigh garment. NMES training will consist of 20-minute stimulation sessions performed concurrently with the exercise program.
  For the BFR training, the automatic Delfi's PTS Personalized Tourniquet System for Blood Flow Restriction (Delfi Medical, Vancouver, BC, Canada) with variable contour nylon cuff (11.5 cm × 86 cm, 2.5 mm thick) will be used. The Delfi PTS system automatically adjusts pressure around the set occlusion pressure. The Low BFR group will have the pressure set at 20 mmHg.
  Interventions: Device: NMES and exercise supplemented with low BFR

INTERVENTIONS:
Device: NMES and exercise supplemented with high BFR — The BFR-NMES-Exercise training consists of 20-min sessions performed concurrently with NMES and exercise in the clinic 2x a week for a total of 18 in-clinic sessions. Using the Delfi PTS Personalized Tourniquet System for Blood Flow Restriction at 80% of LOP, the participant performs 4 exercise sets of 60 repetitions (5 seconds ea) for 5 minutes, with a 1-minute BFR deflation between sets. The standard exercise rehabilitation protocol for PFPS combines open chain and closed chain quadriceps strengthening exercises: active straight leg raises, quadriceps straightening, step up, and squats. NMES training consists of 20-minute sessions: a 2-min warm-up, 15-min work-out, and a 3-min cool down using the KneeHAB® XP "Multipath" stimulation system which changes the current pathways between the electrodes for preset periods within each pulse, allowing for higher stimulation intensities that maximizes muscle fibre recruitment and minimizes muscle fatigue.
  Arms: NMES and exercise supplemented with high BFR
Device: NMES and exercise supplemented with low BFR — The BFR-NMES-Exercise training consists of 20-min sessions performed concurrently with NMES and exercise in the clinic 2x a week for a total of 18 in-clinic sessions. Using the Delfi PTS Personalized Tourniquet System for Blood Flow Restriction at 20mmHG venous pressure (no blood flow restricted), the participant performs 4 exercise sets of 60 repetitions (5 seconds ea) for 5 minutes, with a 1-minute BFR deflation between sets. The standard exercise rehabilitation protocol for PFPS combines open chain and closed chain quadriceps strengthening exercises: active straight leg raises, quadriceps straightening, step up, and squats. NMES training consists of 20-minute sessions: a 2-min warm-up, 15-min work-out, and a 3-min cool down using the KneeHAB® XP "Multipath" stimulation system which changes the current pathways between the electrodes for preset periods within each pulse, allowing for higher stimulation intensities that maximizes muscle fibre recruitment and minimizes muscle fatigue.
  Arms: NMES and exercise supplemented with low BFR

SUMMARY:
The overall objective of this project is to compare two self-managed treatment regimens for PFPS: (1) NMES-Exercise supplemented with high BFR LOP of 80% and (2) NMES Exercise augmented with a low percentage of BFR LOP at 20 mmHG (BFR-sham). Each of the two treatment arms will perform a fixed exercise protocol singularly and in combination with BFR-NMES, and NMES alone. The specific aims of the study are 1) To determine whether self-managed NMES-Exercise program supplemented with a high BFR of 80% LOP (limb occlusion pressure) is significantly more efficacious than NMES-Exercise with low BFR LOP set at 20 mmHG (sham) in improving muscle strength of the lower extremity, daily physical activity and mobility; and 2) To determine whether NMES-Exercise with high LOP BFR therapy improves QOL and PFPS symptoms significantly more than NMES-Exercise with low LOP BFR.

DETAILED DESCRIPTION:
The long-term goal is to identify effective self-managed therapies for military members that will return them to duty as quickly as possible. The overall objective of this project is to compare two self-managed treatment regimens for PFPS: (1) NMES-Exercise supplemented with high BFR LOP of 80% and (2) NMESExercise augmented with a low percentage of BFR LOP at 20 mmHG (BFR-sham). Each of the two treatment arms will perform a fixed exercise protocol singularly and in combination with BFR-NMES, and NMES alone.

The rationale for this study is that by limiting blood flow to an exercising limb using both active and passive exercise is expected to significantly improve lower extremity muscle strength, mobility, quality of life (QOL) and pain. The central hypothesis is that the combination of NMES/exercise of the injured leg supplemented with BFR set at 80% LOP will show significantly greater improvements in muscle strength, mobility, pain, daily activity and QOL than the NMES-Exercise with BFR set at a very low percentage of LOP at 20 mmHG. To test this hypothesis, the investigators will address the following specific aims:

a1. To determine whether self-managed NMES-Exercise program supplemented with a high BFR of 80% LOP (limb occlusion pressure) is significantly more efficacious than NMES-Exercise with low BFR LOP set at 20 mmHG (sham) in improving muscle strength of the lower extremity, daily physical activity and mobility. Muscle strength will be measured by isometric peak torque of the left and right knee and hip posterolateral stabilizers; physical activity will be measured by steps walked and energy (kcal) expenditure/day; and mobility by time to complete a stair climb, step down test, distance walked in 6 minutes, and number of times to complete the chair rise.

a2. To determine whether NMES-Exercise with high LOP BFR therapy improves QOL and PFPS symptoms significantly more than NMES-Exercise with low LOP BFR. QOL will be measured by the SF-12 Health Survey and the Center for Epidemiological Studies-Depression (CES-D) scale. Symptoms of PFPS will be quantified by the Anterior Knee Pain Scale and IKDC subjective knee form.

The investigators expect to demonstrate that these combined multimodality therapies of a self-managed NMES-Exercise program supplemented with high (80%) LOP BFR-NMES-Exercise is more efficacious than a low percentage of LOP BFR-NMES-Exercise (sham). Positive results will translate into therapy options for PFPS that can be used by health care providers to accelerate rehabilitation, speed return to world-wide duty status, decrease symptoms, and lower medical costs. Moreover, these approaches are safe, easy to use and non-pharmacological.

ELIGIBILITY:
Inclusion Criteria:

- Active duty military personnel who are:

1. diagnosed with knee pain, categorized as anterior or retropatellar in one or both knees;
2. self-reported difficulty performing at least two or more of the following activities associated with knee pain: prolonged sitting, stair climbing, running, jumping, and repetitive movements such as kneeling or squatting or stooping;
3. military service member at the time of diagnosis and length of study;
4. age ≥18 and <45 years; and
5. able to provide freely given informed consent.

Exclusion Criteria:

1. fracture or injury to external knee structures such that knee extension or flexion is impaired;
2. a significant co-morbid medical condition (such as severe hypertension, neurological disorder, sickle cell anemia, or pacemaker/defibrillator) in which BFR, NMES strength training, or unsupervised exercise is contraindicated and would pose a safety threat or impair ability to participate;
3. previous knee surgeries (i.e., tibiofemoral, patellofemoral) excluding knee arthroscopy > 3 years;
4. knee instability or recurrent patella dislocation or subluxation;
5. inability or unwillingness to participate in an exercise or strengthening program;
6. reduced sensory perception in the lower extremities;
7. pregnancy;
8. Any vascular disorder (varicose veins, Hx of DVT); or
9. unwillingness to accept random assignment.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Lower Extremity Muscle Strength- Extension | Time Frame: 9 weeks
  Strength of knee extension muscle groups will be measured using the Nicholas Manual Muscle Tester (NMMT). The participant will be positioned with a small towel roll placed distally to support the femur in 90-degree hip flexion. The participant's knee will be placed in 70º knee flexion using a goniometer. The distance from the tibial tuberosity (TT) to the superior aspect of the medial malleolus will be measured.
  For knee extension, the first measurement will be taken using standard NMMT protocol (0.6 X the distance from the tibial tuberosity to the superior aspect of the medial malleolus). Participants will perform three maximal efforts holding contractions for 4 seconds, separated by 30-sec rest; the highest value of the will be accepted (kg).
Change in Lower Extremity Muscle Strength- Flexion | Time Frame: 9 weeks
  Strength of knee flexion muscle groups will be measured using the Nicholas Manual Muscle Tester (NMMT). The participant will be positioned with a small towel roll placed distally to support the femur in 90-degree hip flexion. The participant's knee will be placed in 70º knee flexion using a goniometer. The distance from the tibial tuberosity (TT) to the superior aspect of the medial malleolus will be measured.
  For knee flexion, the NMMT will be positioned 0.6X distance from TT to superior border of medial malleolus on the dorsal limb side. Participants will perform three maximal efforts holding contractions for 4 seconds, separated by 30-sec rest; the highest value of the will be accepted (kg).
Change in Lower Extremity Muscle Strength- Hip Posterolateral Stabilizer | Time Frame: 9 weeks
  Strength of hip posterolateral stabilizer muscle groups will be measured using the Nicholas Manual Muscle Tester (NMMT). The hip stability isometric test (HipSIT) will be measured using the NMMT as described by Almeida et al. Participants will perform three maximal efforts holding contractions for 4 seconds, separated by 30-sec rest; the highest value of the will be accepted (kg).
Change in Mobility- Timed Stair Climb Test | Time Frame: 9 weeks
  Tests the activity of stair climbing. The test will begin with participants ascending up four steps (6-inch rise, 11.5-inch run) to a 30-inch square platform, and then descending to the bottom of the stairs. Participants will climb the stairs at a self-selected pace using the handrails if necessary.
  Each participant will complete two complete rounds, if possible, and the two times will be averaged to produce one score.
Change in Mobility- Forward Step-Down Test | Time Frame: 9 weeks
  This is a specific function test for PFPS, putting weight bearing stress during a movement that mimics stair descent. The test is performed from a 20 cm (8 inch) high platform. The participant steps forward and down toward the floor from a single-leg stance with a straight knee (hands on hips). The knee of the stance leg bends until the opposite foot lightly touches the floor with the heel and then returns to full knee extension. The heel touching the floor is not to be used to accelerate back onto the platform. This counts as one repetition; the number of repetitions performed in 30 seconds is recorded. Both legs are tested separately.
Change in Mobility- 30-Second Chair Stand Test | Time Frame: 9 weeks
  This assesses lower-body strength mimicking squatting. The participant completes as many full stands as possible in 30 seconds. The participant sits in the middle of the chair, feet flat on the floor with arms crossed at the wrists and held against the chest. When instructed, the participant rises to a full stand, and then returns to a fully seated position. The number of completed rises will be recorded.
Change in Mobility- 6-Minute Walk Test | Time Frame: 9 weeks
  This is a submaximal test of functional capacity and measures the distance a participant walks at a "fast" pace over a 6-minute period. Participants will "walk as quickly as you can" with the opportunity to stop and rest if required. This test measures functional capacity of walking.
Change in Physical Activity- Steps walked | Time Frame: 9 weeks
  Physical activity will be measured using the Fitbit Charge (San Francisco, CA). The Charge is a wrist-worn, three-axis accelerometer that measures steps walked, distance traveled, energy expenditure and floors climbed. Steps walked will be assessed as the number of steps walked in 24 hours.
  Baseline data will be ascertained by wearing the Charge for 3 days while maintaining a typical activity pattern. Subsequently, the device will be worn daily for 9 weeks.
Change in Physical Activity- Energy expenditure | Time Frame: 9 weeks
  Physical activity will be measured using the Fitbit Charge (San Francisco, CA). The Charge is a wrist-worn, three-axis accelerometer that measures steps walked, distance traveled, energy expenditure and floors climbed. Energy expenditure will be assessed as the calories expended in 24 hours.
  Baseline data will be ascertained by wearing the Charge for 3 days while maintaining a typical activity pattern. Subsequently, the device will be worn daily for 9 weeks.

SECONDARY OUTCOMES:
Change in Symptoms of PFPS- Knee pain limiting actiivty (AKPS) | Time Frame: 9 weeks
  Pain associated with activity limitations will be measured by the Kujala Anterior Knee Pain Scale, a 13-item knee specific self-report questionnaire. Scores range from 0 to 100 with higher scores indicating better performance.
Change in Symptoms of PFPS- Pain at rest and post-activity (VAS) | Time Frame: 9 weeks
  The Visual Analog Scale (VAS) of pain will be used to assess pain at rest and after activity. Participants will complete this scale following the stair climb, step down test, 6-minute walk and the chair rise test. This VAS pain subscale is a 100-mm horizontal line index with descriptive anchors at each end. At the far left (0.0cm) is "no pain" and at the far right (10 cm) is "worst possible pain". The participant is instructed to place a vertical line at some point between the anchors to describe his/her level of pain. The VAS pain scale shows high correlations with acute pain levels.
Change in Symptoms of PFPS- Knee Injury and Disability (IKDC) | Time Frame: 9 weeks
  Knee Injury and disability will be measured by the International Knee Documentation Committee (IKDC) subjective knee form, a well standardized outcomes questionnaire that is knee-specific and assesses patients with various knee disorders. The 18-item instrument assesses symptoms, function and level of sports participation for those with an injured knee.
Change in Quality of Life- Overall: The Short Form Health Survey Version 2.0 (SF-12v2) Health Survey | Time Frame: 9 weeks
  The Short Form Health Survey Version 2.0 (SF-12v2) Health Survey will be used to determine each participant's overall health-related quality of life. The SF12v2 has two summary scores for physical (PCS) and mental health (MCS). Raw scores for each subscale are computed using the scores of 12 questions ranging from 0-100. Zero score indicates the lowest level and 100 indicates the highest level of health. The PCS and MCS subscales are norm-based for different age groups because of the variance in PCS and MCS scores over the life span.

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Talbot, PhD, EdD, RN, Principal Investigator — University of Tennessee Health Sciences Center
Locations (1):
- Blanchfield Army Community Hospital (BACH), Fort Campbell North, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Talbot LA, Webb L, Morrell C, Enochs K, Hillner J, Fagan M, Metter EJ. Electromyostimulation With Blood Flow Restriction for Patellofemoral Pain Syndrome in Active Duty Military Personnel: A Randomized Controlled Trial. Mil Med. 2023 Jul 22;188(7-8):e1859-e1868. doi: 10.1093/milmed/usad029. Epub 2023 Feb 20. PMID 36807977

DOCUMENTS (1):
  • Informed Consent Form (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/15/NCT04086615/ICF_000.pdf